CLINICAL TRIAL: NCT01943539
Title: A Study to Assess the Feasibility of EVO Gameplay to Engage Children With Attention Deficit Hyperactivity Disorder (ADHD) and to Evaluate Cognitive Interference in Children Ages 8 to 12 Years Old With ADHD Compared to Neuro-typical Children
Brief Title: Cognitive ADHD Videogame Exploratory Study
Acronym: CAVES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akili Interactive Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Akili-001
Record Dates: First submitted 2013-09-05; First posted 2013-09-17 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EVO Game Play (Experimental): Neuro-typical controls and ADHD will receive EVO game play.
  Interventions: Device: Neuro-typical controls and ADHD will receive EVO game play.

INTERVENTIONS:
Device: Neuro-typical controls and ADHD will receive EVO game play. — EVO mobile video application

SUMMARY:
A study in ADHD and neuro-typical children to assess EVO game play over 29 days.

DETAILED DESCRIPTION:
A study in children ages 8 to 12 to assess EVO cognitive game play. The study examines two populations, children diagnosed with ADHD (ADHD and not on medication) and neuro-typical children. The investigators plan to evaluate 80 subjects (N = 40 per group) in three site locations over a 29 day study period. The 29 day study period includes 2 in-clinic sessions and 27 days of out-patient game play. During the 27 days of out-patient game play, the subjects will be instructed to play EVO 5 days per week for typically 30 minutes per day

The investigators' hypothesis is that EVO will be playable and interesting to ADHD children and cognitive measures, as captured by EVO, will show a difference between ADHD children and age-matched neuro-typical children.

ELIGIBILITY:
Inclusion Criteria:

1. Age 8 to 12 at the time of parental informed consent.
2. Confirmed ADHD diagnosis at clinic per MINI-Kid (ADHD Cohort)
3. Baseline ADHD-RS-IV score >= 24 (ADHD Cohort), obtained at clinic
4. Baseline ADHD-RS-IV score <=13 (Neuro-typical Cohort), obtained at clinic
5. Consistently off ADHD drug for 1 week. Drugs include: Pre specified, oral psychostimulants (ADDERALL XR® [mixed salts of a single-entity amphetamine product], VYVANSE® [lisdexamfetamine dimesylate], CONCERTA® [methylphenidate HCl], FOCALIN XR® [dexmethylphenidate HCl], RITALIN LA® [methylphenidate HCl extended-release], METADATE CD® [methylphenidate HCl, USP], or FDA-approved generic equivalents )for 1 month (Other than ADHD drud
6. Consistently off Psychotropic drug for 1 month (Other than ADHD drug noted above)
7. Ability to follow written and verbal instructions (English)
8. Girls or Boys (Gender-matched - 30% girls minimum)
9. Functioning at an age-appropriate level intellectually.
10. Ability to comply with all the testing and requirements.

Exclusion Criteria:

1. Current, controlled (requiring a restricted medication) or uncontrolled, comorbid psychiatric diagnosis with significant symptoms such as post-traumatic stress disorder, psychosis, bipolar illness, pervasive developmental disorder, severe obsessive compulsive disorder, severe depressive or severe anxiety disorder, conduct disorder, or other symptomatic manifestations that in the opinion of the Investigator that may confound study data/assessments (per MINI-Kid).
2. Within the last 4 weeks, subject has entered or exited behavioral therapy. The subject should inform the Investigator if they intend to change their behavioral therapy during the 4 weeks of the study.
3. Subject is currently considered a suicide risk in the opinion of the Investigator, has previously made a suicide attempt, or has a prior history of, or is currently demonstrating active suicidal ideation or self-injurious behavior (per C-SSRS).
4. History of failure to respond to an adequate trial of 2 treatments for ADHD (consisting of an appropriate dose and adequate duration of therapy and failure in efficacy in the opinion of the Investigator).
5. Motor condition that prevents game playing
6. Recent history (within the past 6 months) of suspected substance abuse or dependence.
7. History of seizures (exclusive of febrile seizures), a tic disorder, significant tics, or a current diagnosis of Tourette's Disorder.
8. Taken part in a clinical trial within 30 days prior to screening.
9. Diagnosis of color blindness
10. Regular use of psychoactive drugs that in the opinion of the Investigator may confound study data/assessments.
11. Any other medical condition that in the opinion of the Investigator may confound study data/assessments.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2013-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Cutler, MD, Principal Investigator — Florida Clinical Research Center, LLC
Locations (2):
- United States (2):
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Duke University, Durham, North Carolina

REFERENCES:
- [Derived] Davis NO, Bower J, Kollins SH. Proof-of-concept study of an at-home, engaging, digital intervention for pediatric ADHD. PLoS One. 2018 Jan 11;13(1):e0189749. doi: 10.1371/journal.pone.0189749. eCollection 2018. PMID 29324745

RESULTS

PARTICIPANT FLOW:
Groups:
- Neuro-typical Controls: Non-ADHD neuro-typical children
- ADHD: Children diagnosed with ADHD and not on ADHD medication.
Period: Overall Study
Arm/Group | Neuro-typical Controls | ADHD
Started | 44 | 40
Completed | 40 | 40
Not Completed | 4 | 0
Not completed — Non-compliance with at-home intervention | 4 | 0

BASELINE CHARACTERISTICS:
Population: 84 subjects were started, 4 subjects (neurotypical) were excluded from the analysis for non-compliance with the at-home intervention use.
Arm/Group | EVO Game Play
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 40 participants were analyzed in both the ADHD and neuro-typical arms.
  years
    ADHD: number analyzed (Participants) | 40
    ADHD | 10.35 (1.24)
    Neuro-typical: number analyzed (Participants) | 40
    Neuro-typical | 10.54 (1.49)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: 40 participants were analyzed in both the ADHD and neuro-typical arms.
  Participants
    ADHD: number analyzed (Participants) | 40
    ADHD: Female | 16
    ADHD: Male | 24
    Neuro-typical: number analyzed (Participants) | 40
    Neuro-typical: Female | 19
    Neuro-typical: Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 80

OUTCOME MEASURES:

1. Primary Outcome: Reaction Time in EVO Gameplay
Description: EVO employs a perceptual discrimination attention/memory task as well as a continuous visuomotor "driving" task. Subjects were instructed to target a pre-specified stimulus, and ignore all other stimuli while navigating a road-like course. Reaction time was measured as the time between the initial presentation of the pre-specified target and when the subject tapped the tablet screen. Longer reaction times indicated a larger deficit in multitasking.
Time Frame: 28 days
Population: All subjects completing 4 weeks of at-home play and returning to the clinic on DAY 28.
Measure: Mean (Standard Deviation); unit: Reaction time (ms)
Arm/Group | EVO Game Play
Number analyzed (Participants) | 80
Reaction time (ms)
  ADHD: number analyzed (Participants) | 40
  ADHD | 520 (0.091)
  Neuro-typical: number analyzed (Participants) | 40
  Neuro-typical | 480 (0.052)
Statistical Analysis 1: Comparison: EVO Game Play; Test type: Superiority; p = 0.008, t-test, 2 sided; Effect Size = 0.62

2. Primary Outcome: Number of Participants With Non-Treatment Related Adverse Events
Description: Another objective of this study is to evaluate the safety of EVO game play based on treatment-emergent adverse events (TEAEs) that may occur during this 28-day period of time.
Time Frame: Day 0 through Day 28 of the study
Population: All subjects completing 4 weeks of at-home play and returning to the clinic on DAY 28.
Measure: Count of Participants; unit: Participants
Arm/Group | EVO Game Play
Number analyzed (Participants) | 80
Participants
  ADHD (non-treatment related AEs): number analyzed (Participants) | 40
  ADHD (non-treatment related AEs) | 4
  Neuro-typical (non-treatment related AEs): number analyzed (Participants) | 40
  Neuro-typical (non-treatment related AEs) | 5

3. Secondary Outcome: Time Spent Completing the Intervention
Description: Time spent on completing the intervention is based on the prescribed therapy of 800 total minutes, or 13.3 hours, over the course of 28 days (7 sessions of EVO per day for 5 days per week for 4 weeks with each session lasting approximately 5.7 minutes long).
Time Frame: 28 days
Population: All subjects completing 4 weeks of at-home play and returning to the clinic on DAY 28.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | EVO Game Play
Number analyzed (Participants) | 80
Hours
  ADHD: number analyzed (Participants) | 40
  ADHD | 10.8 (2.8)
  Neuro-typical: number analyzed (Participants) | 40
  Neuro-typical | 11.5 (2.6)

4. Other Pre Specified Outcome: Mean of Differences in TOVA Attention Performance Index (API) at Baseline (Day 0) and at Day 28
Description: TOVA API is a comparison of the subject's scores based on selected measures that persons with an independent diagnosis of ADHD frequently demonstrated. The API is calculated from variability, response time, and D' (D Prime) using the following formula:
  API = Response Time Z score (Half 1) + D' Z score (Half 2) + Variability Z score (Total) + 1.80
  where Response Time is the average time it takes to respond correctly to a target, d' (D Prime) score is a response discriminability score reflecting the ratio of hits to "false alarms", and Variability is a measure of consistency of speed of responding based on the standard deviation of the mean correct response times. API tells how similar the score is to the ADHD profile. A score of less than -1.8 indicates that the subject had similar performance to a normative ADHD population. A lower score indicates a more severe ADHD profile.
  The calculation for difference in TOVA API was API at Baseline (Day 0) minus API at Day 28.
Time Frame: Day 0 and Day 28
Population: All subjects completing 4 weeks of at-home play and returning to the clinic on DAY 28.
Measure: Mean (95% Confidence Interval); unit: Cumulative z-score
Groups:
- Neurotypical Controls: Non-ADHD neuro-typical children
- ADHD: Children diagnosed with ADHD and not taking ADHD medication
Arm/Group | Neurotypical Controls | ADHD
Number analyzed (Participants) | 40 | 40
Cumulative z-score | -0.39 [-1.16 to 0.37] | -1.43 [-2.75 to -0.12]

ADVERSE EVENTS:
Time Frame: 8 months
Groups:
- Neurotypical Controls: Non-ADHD neurotypical children
- ADHD: Children diagnosed with ADHD and no on ADHD medication
Arm/Group | Neurotypical Controls | ADHD
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/40
Serious Adverse Events (participants affected / at risk) | 1/44 | 0/40
Other Adverse Events (participants affected / at risk) | 4/44 | 4/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neurotypical Controls (N=44) | ADHD (N=40)
Acute reflux esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neurotypical Controls (N=44) | ADHD (N=40)
Toothache (General disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 2 (2)
Viral gastroenteritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Foot pain (General disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No